CLINICAL TRIAL: NCT01996111
Title: A Prospective, Randomized, Controlled, Blinded, Comparative Study of Dehydrated Human Amnion/Chorion Membrane Micrografts(dHACM) Injectable in the Treatment of Recalcitrant Plantar Fasciitis
Brief Title: Dehydrated Human Amnion/Chorion Membrane Micrografts(dHACM) Injectable in the Treatment of Recalcitrant Plantar Fasciitis
Acronym: dHACM
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Change in Regulatory Status
Sponsor: MiMedx Group, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: AIPF003
Record Dates: First submitted 2013-10-10; First posted 2013-11-27 (Estimated); Last update posted 2014-06-13 (Estimated); Status verified 2014-06

CONDITIONS: Plantar Fasciitis
Keywords: plantar fasciitis
MeSH Terms: conditions — Fasciitis, Plantar | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- • Group 2: (Experimental): Injection of 1.0 cc of 10 mg/ml micrograft dHACM suspension
  Interventions: Procedure: Injection of 1.0 cc of 10 mg/ml micrograft dHACM suspension
- • Group 3: (Experimental): Injection of 1.0 cc of 20 mg/ml micrograft dHACM suspension
  Interventions: Procedure: Injection of 1.0 cc of 20 mg/ml micrograft dHACM suspension
- • Group 4: (Experimental): Injection of 1.0 cc of 40 mg/ml micrograft dHACM suspension
  Interventions: Procedure: Injection of 1.0 cc of 40 mg/ml micrograft dHACM suspension
- • Group 1 (Placebo Comparator): • Injection of 1.0 cc of 0.9% Saline
  Interventions: Procedure: Injection of 1.0 cc of 0.9% Saline

INTERVENTIONS:
Procedure: Injection of 1.0 cc of 0.9% Saline — Injection of 1.0 cc of 0.9% Saline into affected area
  Arms: • Group 1
Procedure: Injection of 1.0 cc of 10 mg/ml micrograft dHACM suspension — Injection of 1.0 cc of 10 mg/ml micrograft dHACM suspension into affected area
  Arms: • Group 2:
Procedure: Injection of 1.0 cc of 20 mg/ml micrograft dHACM suspension — Injection of 1.0 cc of 20 mg/ml micrograft dHACM suspension into affected area
  Arms: • Group 3:
Procedure: Injection of 1.0 cc of 40 mg/ml micrograft dHACM suspension — Injection of 1.0 cc of 40 mg/ml micrograft dHACM suspension into affected area
  Arms: • Group 4:

SUMMARY:
This is a prospective, controlled, randomized, blinded and comparative, single-center clinical trial comparing the improvement of patients with recalcitrant plantar fasciitis symptoms that have received standard of care versus treatment with differing amounts of injectable dehydrated human amnion/chorion membrane micrografts(dHACM).

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years old.
2. Both male and female patients will be selected.
3. Plantar fasciitis has been treated with conservative usual care for at least 8 weeks, including at least three of the following modalities

   * Rest, Ice, Compression, Elevation (RICE)
   * Corticosteroid injection
   * Stretching exercises
   * Non-steroidal Anti-Inflammatory Drugs (NSAIDs)
   * Orthotics
4. Females of childbearing potential must be willing to use acceptable methods of contraception (birth control pills, barriers, or abstinence).
5. Patient understands and is willing to participate in the clinical study and can comply with weekly visits and the follow-up regimen.
6. Patient has read and signed the IRB/IEC approved Informed Consent Form before screening procedures are undertaken.

Exclusion Criteria

1. Prior surgery at the site.
2. Site that exhibits clinical signs and symptoms of infection.
3. History of chronic plantar fasciitis of more than twelve months.
4. Evidence of significant neurological disease of the feet.
5. Non-ambulatory patients.
6. The presence of comorbidities that can be confused with or can exacerbate the condition including:

   * Calcaneal stress fracture
   * Nerve entrapment syndrome (Baxter's Nerve Entrapment or Tarsal Tunnel Syndrome)
   * Plantar fascial rupture
   * Systemic disorders associated with enthesiopathy (such as Gout, Reiter's syndrome, rheumatoid arthritis, etc.)
   * Achilles tendonitis
   * Fat pad atrophy
   * Fibromyalgia
   * Diabetics with neuropathy
7. Patients with a history of more than two weeks treatment with immuno-suppressants (including systemic corticosteroids), cytotoxic chemotherapy within one month prior to initial screening, or who receive such medications during the screening period, or who are anticipated to require such medications during the course of the study.
8. Patients on any investigational drug(s) or therapeutic device(s) within 30 days preceding screening.
9. History of radiation therapy at the site.
10. Known history of having Acquired Immunodeficiency Syndrome (AIDS) or HIV.
11. Study foot has been previously treated with tissue engineered materials within the last 30 days.
12. Patients who are unable to understand the aims and objectives of the trial.
13. Presence of any condition(s) which seriously compromises the subject's ability to complete this study, or has a known history of poor adherence with medical treatment.
14. Pregnant or breast feeding. No pregnancy within the past 6 months.
15. Allergy to Gentamicin and/or Streptomycin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2013-09; Primary Completion 2014-03 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Reduction of inflammation as measured by AOFAS Hindfoot scores | 8 Weeks
  The primary objective of this study is to compare the efficacy of the different treatment amounts in reduction of inflammation as measured by AOFAS Hindfoot scores.

SECONDARY OUTCOMES:
Return to normal activities more quickly than with standard of care | 8 Weeks
  The secondary objective is to demonstrate that patients treated with micronized dHACM injectable will return to normal activities more quickly than with standard of care.
Pain as measured by 0-10 Numeric Rating Scale | 12 weeks
  Patient pain scores will be assessed between all groups.

OTHER OUTCOMES:
Quality of Life as measured by SF-36 | 8 weeks
  SF-36 scores between all groups before and after treatment over a period of eight weeks. Physical Component Score (PCS) and Mental Component Score (MCS) will be evaluation at 8 weeks and compared to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Charles M. Zelen, DPM, Principal Investigator — Professional Education and Research Institute
Locations (1):
- Professional Education and Research Institute, Roanoke, Virginia, United States